CLINICAL TRIAL: NCT00975117
Title: Assessment of the Efficacy of Dietary Supplement Spermotrend in the Treatment of Male Infertility
Brief Title: Spermotrend in the Treatment of Male Infertility
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Miguel Aguilar Charara, "Ramón González Coro" Gynecologic and Obstetric Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAT-0905-CU
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Male Infertility
Keywords: Dietary supplement; male infertility; spermatogenesis
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Spermotrend (Experimental)
  Interventions: Dietary Supplement: Spermotrend

INTERVENTIONS:
Dietary Supplement: Placebo — One Placebo tablet (Orally administered) twice a day, for 12 weeks.
  Arms: Placebo
Dietary Supplement: Spermotrend — One Spermotrend tablet (Orally administered) twice a day, for 12 weeks
  Arms: Spermotrend

SUMMARY:
The purpose of this study is to determine whether the administration of the dietary supplement Spermotrend improves spermatogenesis parameters in subjects with male infertility unrelated to major testicular conditions. The duration of this double-blind placebo controlled phase 3 clinical trial will be 24 weeks. The estimated number of males with infertility to be recruited and randomized for the study is 86.

ELIGIBILITY:
Inclusion Criteria:

* Male infertility unrelated to major testicular conditions
* Must have at least one altered seminal parameter.
* Signed informed consent

Exclusion Criteria:

* Hydrocele, varicocele, orchitis, epididymitis, irradiation or Chemotherapy.
* Previously treated and cured testicular condition.
* Non-transmissible chronic diseases
* Use of antioxidant agents within 6 months.
* Use of vitamins within 6 months.
* Use of anti-inflammatory drugs within 6 months.
* Use of hormones prescribed by an andrologist within 6 months
* Positive serology/HIV
* Leukocytospermia

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Parameters of seminal analysis at weeks 24 | 24 weeks

SECONDARY OUTCOMES:
Fertilization achievement | 24 weeks
Presence of mild or severe adverse effects | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Aguilar Charara, MD, Principal Investigator — "Ramón González Coro" Gynecologic and Obstetric Hospital
Locations (1):
- "Ramón González Coro" Gynecologic and Obstetric Hospital, Havana, La Habana, Cuba

REFERENCES:
- [Derived] de Ligny W, Smits RM, Mackenzie-Proctor R, Jordan V, Fleischer K, de Bruin JP, Showell MG. Antioxidants for male subfertility. Cochrane Database Syst Rev. 2022 May 4;5(5):CD007411. doi: 10.1002/14651858.CD007411.pub5. PMID 35506389